CLINICAL TRIAL: NCT00408551
Title: A Phase II Multi-Institutional Efficacy and Safety Study of Chemotherapy With Selective Internal Radiation Treatment Using Y-90 Microspheres (CHEMO-SIRT) in Patients With Colorectal Cancer Liver Metastasis
Brief Title: Chemotherapy and Internal Radiation in Treating Patients With Colorectal Cancer That Has Spread to the Liver
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goshen Health System (Other)
Responsible Party: Kenneth Lee Pennington, Center for Cancer Care at Goshen General Hospital
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000515900; CCCGHS-CHEMO-SIRT
Record Dates: First submitted 2006-12-06; First posted 2006-12-07 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; liver metastases; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Floxuridine; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

ARMS (3):
- FOLFOX6 (Experimental): Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continously over 46 hours beginning on day 1.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin
- FOLFIRI (Experimental): Patients receive irinotecan hydrochloride IV over 1 hour and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1.
  Interventions: Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium
- FUDR (Experimental): Patients receive floxuridine IV continuously on days 1-14.
  Interventions: Drug: floxuridine

INTERVENTIONS:
Drug: floxuridine — Given IV
  Arms: FUDR
Drug: fluorouracil — Given IV
  Arms: FOLFIRI; FOLFOX6
Drug: irinotecan hydrochloride — Given IV
  Arms: FOLFIRI
Drug: leucovorin calcium — Given IV
  Arms: FOLFIRI; FOLFOX6
Drug: oxaliplatin — Given IV
  Arms: FOLFOX6

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving chemotherapy together with internal radiation may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving chemotherapy together with internal radiation works in treating patients with colorectal cancer that has spread to the liver.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the tumor response, as measured by total tumor mass, carcinoembryonic antigen (CEA) level, measurable tumor volume by CT scan, and metabolic response by positron emission tomography (PET) scan, in patients with colorectal cancer metastatic to the liver undergoing chemotherapy and selective internal radiation therapy (SIRT) comprising yttrium Y 90 resin microspheres.
* Evaluate the hepatic toxicity of this regimen, as measured by ALT, alkaline phosphatase, and bilirubin levels, in these patients.

Secondary

* Evaluate the therapeutic efficacy of this regimen, using time to in-liver disease progression as an end point, in these patients.
* Evaluate the therapeutic efficacy of this regimen, using down-staging to resectability as an end point, in these patients.

OUTLINE: This is a multicenter study.

Patients receive 1 of the following chemotherapy regimens:

* FOLFOX6: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continously over 46 hours beginning on day 1.
* FOLFIRI: Patients receive irinotecan hydrochloride IV over 1 hour and leucovorin calcium IV over 2 hours on day 1. Patients also receive fluorouracil IV continuously over 46 hours beginning on day 1.
* FUDR: Patients receive floxuridine IV continuously on days 1-14. In all chemotherapy regimens, treatment repeats every 2 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients also undergo selective internal radiation therapy (SIRT) comprising yttrium Y 90 resin microspheres on day 2 of chemotherapy course 1 (for patients receiving FOLFOX6 or FOLFIRI chemotherapy regimens) or on day 1, 2, 3, 4, or 5 of course 1 (for patients receiving FUDR chemotherapy regimen). SIRT may repeat in week 10 or 12.

In week 18, patients may undergo surgery if down-staging has occurred or they may receive more chemotherapy.

After completion of study therapy, patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer* meeting 1 of the following criteria:

  * Metachronous metastasis after resection of Dukes A-C (i.e., stage I-III) primary colon cancer with or without adjuvant chemotherapy
  * Metachronous metastasis after resection of primary rectal cancer with neoadjuvant or adjuvant chemotherapy
  * Synchronous metastatic liver disease with symptomatic or asymptomatic primary colorectal cancer NOTE: *If the patient has a second malignancy with liver metastasis potential, histologic or cytologic confirmation of the liver lesions may be performed as clinically indicated
* Liver-only or liver-predominant disease with any of the following:

  * Unresected primary disease
  * Limited bone or lung disease
  * Potentially resectable nodal disease
  * Anastomotic disease
* No active CNS metastasis or diffuse peritoneal metastasis
* No hepatic metastases from a second malignancy
* No predominant extrahepatic disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* WBC ≥ 1,500/mm^3
* Creatinine ≤ 2 mg/dL
* Bilirubin ≤ 2 mg/dL (without extrahepatic biliary obstruction)
* Albumin > 2 g/dL
* INR < 1.5 (without anticoagulation)
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior external-beam radiotherapy to the liver
* Concurrent targeted therapy agents (e.g., bevacizumab or cetuximab) allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Tumor response as measured by carcinoembryonic antigen (CEA) level, RECIST criteria, and positron emission tomography (PET) scan
Hepatic toxicity

SECONDARY OUTCOMES:
Therapeutic efficacy based on time from selective internal radiation therapy (SIRT) to in-liver disease progression
Therapeutic efficacy based on the proportion of patients who achieve down-staging among all chemo-SIRT treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L. Pennington, MD, Study Chair — Goshen Health System
Locations (1):
- Center for Cancer Care at Goshen General Hospital, Goshen, Indiana, United States